CLINICAL TRIAL: NCT01986686
Title: Should Elective Resection Follow Nonoperative Management of First Episode of Diverticulitis of the Colon With Abscess and/or Extraluminal Air? A Randomized Controlled Trial.
Brief Title: Recurrence Following Nonoperative Management of 1st Episode of Hinchey II Diverticulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RCB1956
Record Dates: First submitted 2013-08-09; First posted 2013-11-18 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-05

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observational (No Intervention): The observation group will be followed clinically with no further intervention until the primary endpoint is reached.
- Surgery (Active Comparator): The surgery group will be offered colon resection.
  Interventions: Procedure: Colon resection

INTERVENTIONS:
Procedure: Colon resection — Elective robotic/laparoscopic/open colon resection for diverticular disease.
  Arms: Surgery

SUMMARY:
Patients will agree to be randomized to either surgery or observation following nonoperative management of a first episode of Hinchey II diverticulitis. Information will be collected on recurrence rates and major complications in both groups.

DETAILED DESCRIPTION:
This study will randomize patients with first episode of acute diverticulitis of the colon with extraluminal air and/or abscess as defined by CT scan following nonoperative management (NPO, IV antibiotics, percutaneous drainage, and TPN followed by colonoscopy) to observation or elective resection. The primary endpoint is recurrent diverticulitis of the colon defined as an acute episode confirmed at CT scan and requiring hospitalization with IV antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* older than or equal to 18
* history of resolved first episode of diverticulitis with abscess (Hinchey class II) who were successfully treated by our standard protocol
* the diagnosis confirmed by colonoscopy
* Signed informed consent

Exclusion Criteria:

* Prior episode of diverticulitis
* Right sided diverticulitis
* Failure of recovery from first episode, defined as recurrence within one month.
* Cancer found at the site on screening colonoscopy
* Comorbidities prohibiting surgery (as measured by colorectal POSSUM score)
* Immunosuppressed patients
* Hinchey I, III, or IV (diverticulitis with peritonitis and/or free air under the diaphragm)
* Patients who are unable to sign the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-10; Primary Completion 2016-07-16 (Actual); Study Completion 2016-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto C Bergamaschi, MD, PhD, Principal Investigator — Stonybrook University
Locations (1):
- Stony Brook Medicine, Stony Brook, New York, United States

REFERENCES:
- [Derived] You K, Bendl R, Taut C, Sullivan R, Gachabayov M, Bergamaschi R; Study Group on Diverticulitis. Randomized clinical trial of elective resection versus observation in diverticulitis with extraluminal air or abscess initially managed conservatively. Br J Surg. 2018 Jul;105(8):971-979. doi: 10.1002/bjs.10868. Epub 2018 Apr 23. PMID 29683483

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational | Surgery
Started | 81 | 26
Completed | 81 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observational | Surgery | Total
Number analyzed (Participants) | 81 | 26 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.22 (13.05) | 53.31 (13.51) | 54.61 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 11 | 41
  Male | 51 | 15 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Primary Study Endpoint
Description: The primary outcome measure is recurrent diverticulitis of the colon defined as an acute episode confirmed at CT scan and requiring hospitalization with IV antibiotics.
Time Frame: Minimum of 1 year after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Surgery
Number analyzed (Participants) | 81 | 26
Participants | 26 | 2

2. Secondary Outcome: Measure Length of Hospital Stay for Surgery vs Non Surgery Patients
Description: Data collected will include length of hospital stay from the date of admission to discharge day for nonoperative management of the first episode of Hinchey II diverticulitis.
Time Frame: 4 years
Reporting Status: Not Posted

3. Secondary Outcome: Mortality
Description: Data will be collected on percent of patients who die during the follow-up period after enrollment.
Time Frame: 4 years
Reporting Status: Not Posted

4. Secondary Outcome: Readmission
Description: Data will be collected on percent of patients who are readmitted for recurrence or postoperative complications during the follow-up period after enrollment.
Time Frame: 30 days
Reporting Status: Not Posted

5. Secondary Outcome: Post Operative Complications
Description: Data will be collected on percent and type of complications for the surgery arm.
Time Frame: 30 days
Reporting Status: Not Posted

6. Secondary Outcome: Recurrence and Treatment
Description: Data will be collected on recurrence and treatment for recurrent diverticulitis
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Observational | Surgery
Serious Adverse Events (participants affected / at risk) | 0/81 | 2/26
Other Adverse Events (participants affected / at risk) | 0/81 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (N=81) | Surgery (N=26)
Partial small bowel obstruction due to ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Surgical site infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No